CLINICAL TRIAL: NCT06210815
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, and Pharmacokinetic Characteristics of HLX42 (Anti-EGFR ADC) in Patients With Advanced/Metastatic Solid Tumors
Brief Title: A Study of HLX42 in Advanced/Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HLX42-FIH101
Record Dates: First submitted 2024-01-08; First posted 2024-01-18 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Solid Tumor and NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- HLX42 (Experimental): Patients with good tolerability and well controlled disease will receive the treatment once every 3 weeks (Q3W), until progressive disease (PD) without any clinical benefit, initiation of other anti-tumor therapies, death, intolerable toxicity, or withdraw the informed consent (whichever occurs first).
  Interventions: Drug: HLX42

INTERVENTIONS:
Drug: HLX42 — HLX42 is an anti-EGFR monoclonal antibody conjugated with a novel high potency DNA topoisomerase I (topo I) inhibitor, with a drug-antibody-ratio (DAR) of 8.
  Other Names: Anti-EGFR ADC

SUMMARY:
This study is an open-label first-in-human phase I clinical study to evaluate the safety and tolerability of HLX42.

DETAILED DESCRIPTION:
The first stage: This study is an open-label first-in-human phase I clinical study to evaluate the safety and tolerability of HLX42 with escalated doses in the treatment of patients with advanced/metastatic solid tumors. In this study, a 3 + 3 dose escalation method will be adopted, and the patients will be administered with HLX42 at different doses via intravenous infusion. The DLT observation period lasts for 3 weeks after the first administration of HLX42.

The second stage: This is a randimazation, open label, 2 arms, muticentral clinical study, about 30 patients in each arm, the total sample size is about 60. Eligible subjects will be randomized in a 1:1 ratio: Group A: HLX42 2.5 mg/kg; Group B: HLX42 2.0 mg/kg. Stratification: tumor tissue type(adenocarcinoma or squamous carcinoma), EGFR-sensitive mutation status (mutant or wild-type or missing).

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years and ≤ 75 years at the time of signing the ICF, male or female;
2. Patients with histologically or cytologically confirmed advanced/metastatic malignant solid tumors, who are refractory to or intolerable with standard treatment, or for which no standard treatment is available(stage 1); Patients with histologically or cytologically confirmed advanced/metastatic malignant NSCLC, who are refractory to or intolerable with standard treatment, or for which no standard treatment is available(stage 2);
3. At least one measurable lesion as per RECIST 1.1；
4. An ECOG performance status score of 0-1；
5. Life expectancy > 3 months;
6. Adequate organ functions as confirmed by laboratory tests within 7 days prior to the first administration of the investigational product;
7. For patients with hepatocellular carcinoma, Child-Pugh score must be A;

Exclusion Criteria:

1. History of other malignant tumors within 2 years prior to the first administration, except for cured cervical carcinoma in situ or cutaneous basal cell carcinoma;
2. The histopathological type is large cell carcinoma, adenosquamous carcinoma, other types (including but not limited to sarcomatoid carcinoma, lymphoepithelioma-like carcinoma, NUT carcinoma, etc.), or contains neuroendocrine pathological components, etc. (stage 2)；
3. History of (non-infectious) ILD requiring the use of steroids, current ILD, or suspected ILD that cannot be ruled out by imaging at screening;
4. Subjects who are allergic to protein preparations/ monoclonal antibodies/ any component in the formulation of the investigational product;
5. Subjects with known previous serious eye disorders;
6. Active systemic infectious diseases requiring intravenous antibiotics within 2 weeks prior to the first administration of the investigational product;
7. Any poorly-controlled cardiovascular and cerebrovascular clinical symptoms or diseases;
8. Patients who have been assessed as unsuitable for inclusion by the investigator, due to brain metastases, spinal cord compression, or cancerous meningitis with clinical symptoms, or uncontrolled brain or spinal cord metastases that have been evidenced;
9. Patients who have received long-term systemic steroids treatment (equivalent to prednisone > 10 mg/day) or immunosuppressive agents of any other forms, which should be discontinued at least 2 weeks prior to the first infusion of the investigational product;
10. Patients who have used potent CYP2D6/CYP3A inhibitors or inducers within 2 weeks prior to the first administration;
11. Patients who have history of immunodeficiency, including HIV infection or other acquired or congenital immunodeficiencies, or history of organ transplantation;
12. Patients with active HBV or HCV infection or HBV/HCV co-infection;
13. Pregnant or lactating women;
14. Subjects who are not suitable for participating in this clinical study due to any clinical or laboratory abnormalities or other reasons as assessed by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2024-03-14 (Actual); Primary Completion 2026-09-02 (Estimated); Study Completion 2027-06-14 (Estimated)

PRIMARY OUTCOMES:
The Dose-Limiting Toxicity (DLT) of HLX42 within 21 days after the first Administration | From first dose to the end of Cycle 1 (each cycle is 3 weeks).
  DLT refers to the AEs that are determined to be related to the investigational product by the investigator, whose severity will affect the escalation of dose level. In this study, the DLT observation period lasts for 21 days after the first administration of HLX42.
The maximum tolerated dose (MTD) of HLX42 | From first dose to the end of Cycle 1 (each cycle is 3 weeks)
  The highest dose level, at which DLT is observed in no more than one of 6 evaluable patients, is defined as MTD of HLX42.

SECONDARY OUTCOMES:
Objective response rate (ORR) | approximately up to 24 months
  Percentage of participants with complete response (CR) and partial response (PR) based on investigator assessment.
Duration of response (DOR) | approximately up to 24 months.
  Length of time response continued based on investigator's assessment.
Progression-free survival (PFS) | up to approximately up to 24 months
  The PFS is defined as the time from the date of enrollment to the date of the first objective documentation of disease progression (as per RECIST v1.1) or death due to any cause,whichever occurred first.
Overall survival (OS) | approximately up to 24 months
  Time from the date of enrollment to the date of death for any cause.
Cmax | Up to 21 days after the first dose
  Maximum serum concentration (Cmax) of HLX42.
Tmax | Up to 21 days after the first dose
  Time to maximum serum concentration (Tmax) of HLX42.
T1/2 | Up to 21 days after the first dose
  Half-life (T1/2) of HLX42.
ADA (anti-drug antibody) | approximately up to 24 months
  Incidence and titer of ADA of HLX42.
Nab (neutralizing antibody) | approximately up to 24 months
  Incidence and titer of Nab of HLX42.
Number of subjects experiencing adverse events | Day 1 through 90 days after last dose.
  Frequency and seriousness of treatment emergent adverse events (TEAEs).

CONTACTS AND LOCATIONS:
Overall Officials: Yilong Wu, Dr., Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong Provincial People's Hospital, Guangdong, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No